CLINICAL TRIAL: NCT04383249
Title: Routine Pathological Examination of Hernia Sac; Is it a Workload or Necessary?
Status: Completed | Type: Observational
Sponsor: Dr. Ersin Arslan Education and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Uylas, Specialist, Dr. Ersin Arslan Education and Training Hospital
Other Study IDs: 07052020
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Pathology
Keywords: Hernia sac; inguinal hernia; incisional hernia; intestine; omentum
MeSH Terms: conditions — Hernia, Inguinal; Incisional Hernia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pathology result: Pathology result of the hernia sac
  Interventions: Diagnostic Test: Pathology result

INTERVENTIONS:
Diagnostic Test: Pathology result — Pathology result of the hernia sac

SUMMARY:
Routine microscopic examination of the hernia sac is controversial. While some centers do not recommend a routine microscopic examination in inguinal hernias in adult patients, they recommend them in abdominal wall hernias. The investigators aimed to discuss the pathology results and unexpected histopathological findings who underwent abdominal wall and inguinal hernia operation in the light of the literature.

DETAILED DESCRIPTION:
The hernia is defined as the passage of an organ or tissue from one anatomical region to another. Hernia sacs are sent to the pathology department, although there is a difference between clinics. Routine microscopic examination of the hernia sac is controversial. While some centers do not recommend a routine microscopic examination in inguinal hernias in adult patients, they recommend them in abdominal wall hernias. Here, the investigators aimed to discuss the pathology results and unexpected histopathological findings who underwent abdominal wall and inguinal hernia operation in the light of the literature. Patients who have operated hernia and sent hernia sac for histopathological examination were retrospectively screened. Emergency and elective operated patients were included. Hernia repairs without pathology were excluded from the study. Patients' gender, age, operation notes, and pathology results were analyzed. Pathology results were analyzed in two groups as expected findings and unexpected findings. In our study, the probability of encountering an unexpected pathological result was found to be quite low in the pathological evaluation of the hernia sac. Although it may cause additional workload and cost, all hernia sacs should be sent to routine pathological examination. The investigators believe that making savings in these areas through further investigation after the decision of the pathologist.

ELIGIBILITY:
Inclusion Criteria:

* Emergency operated patients
* Elective operated patients

Exclusion Criteria:

* Hernia repairs without pathology examinations

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have operated hernia and sent hernia sac for histopathological examination.
Sampling Method: Non-Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
unexpected finding | 2 or 3 week
  rate of unexpected result

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Ersin Arslan Training and Resource Hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No